CLINICAL TRIAL: NCT00686179
Title: A Double-Blind, Randomised, Multicentre, Placebo-Controlled, 4-Ways Crossover Study to Investigate the Effect on the QT/QTc Interval of Repeated and Escalating Doses of AZD3480 During 6 Days, Using Moxifloxacin as a Positive Control, in Healthy Male Volunteers, CYP2D6 Extensive and Poor Metabolisers.
Brief Title: Investigate the Effect on the QT/QTc Interval of Repeated and Escalating Doses of AZD3480 During 6 Days
Acronym: TQT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans-Göran Hårdemark, MD, PhD, Medical Science Director, AZD3480, AstraZeneca R&D, Södertälje, Sweden
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: D3690C00004; EUdract NO 2007-004859-11
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Healthy
Keywords: TQT; ECG; QT; QTc; AZD3480; ECG(QTc effects)
MeSH Terms: interventions — ispronicline; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Escalating doses of AZD3480 during 6 days
  Interventions: Drug: AZD3480
- 2 (Experimental): Repeated doses of AZD3480 during 6 days
  Interventions: Drug: AZD3480
- 3 (Placebo Comparator): Placebo during 6 days
  Interventions: Drug: PLACEBO
- 4 (Active Comparator): Placebo during 5 days, active day 6
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: AZD3480 — Capsule, oral, single dose, 6 days
  Other Names: TC-1734-226
  Arms: 1; 2
Drug: Moxifloxacin — Capsule(encapsulated), oral, single dose
  Arms: 4
Drug: PLACEBO — Capsule, oral, single dose
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effects on cardiac repolarisation of supratherapeutic doses of AZD3480 compared to placebo in healthy male volunteers, subgrouped as extensive metabolisers and poor metabolisers according to CYP2D6 metabolic capacity, using moxifloxacin as positive control.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a previous study for genotyping for identification to be extensive or poor metaboliser (CYP2D6 enzyme)
* Physically and mentally healthy male volunteers

Exclusion Criteria:

* History of clinically significant diseases or illness.
* Participation in another study the last 3 months
* Prescribed or non-prescribed medications from 3 weeks prior to first treatment day until follow-up except for paracetamol (max 1.5 g per day.)

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
QTcX interval (supratherapeutic doses in comparison to placebo).Subject-specific correction of QT, QTcF and QTcB (supportive outcome variables).Bazett QTcB=QT*RR-1/2Fridericia QTcF=QT'RR-1/3 | 11 dECG measurements x 4 (4-way crossover)

SECONDARY OUTCOMES:
QTcX (therapeutic doses in comparison to placebo).PR-, QRS-, RR-intervals | 11 dECG measurements x 4 (4-way crossover)
Plasma concentration (AUC, Cmax, tmax etc) | 11 PK-measurements x 4 (4-way crossover)
Registration of AEs, blood pressure, ECG, clinical laboratory tests | From enrolment to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Göran Hårdemark, Study Director — Clinical Neuroscience TA AstraZeneca R&D Södertälje, Sweden